CLINICAL TRIAL: NCT05747963
Title: A Prospective, Multicenter, Randomized Clinical Trial for Evaluating the Safety and Efficacy of Software-delivered Cognitive Behavioral Therapy for Insomnia in Patients With Insomnia Disorder.
Brief Title: Software-delivered CBT-I for Insomnia Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Collaborators: Shenzhen Zeen Health Technology Co., Ltd. (Unknown); Peking University First Hospital (Other); Sichuan Provincial People's Hospital (Other); The Second Affiliated Hospital of AFMU (Unknown); Shenzhen Kangning Hospital (Other)
Responsible Party: Principal Investigator, Hongqiang Sun, Professor, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-65
Record Dates: First submitted 2023-02-11; First posted 2023-02-28 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Insomnia Disorder
Keywords: Insomnia Disorder; Software-delivered CBT-I; Randomised Clinical Trial; Digital Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, parallel, randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- software-delivered CBT-I (Experimental): Subjects in intervention group will receive a digital CBT-I for 6 weeks. The automated software incorporates all core elements of CBT-I, tailoring content based on each participant's reported baseline sleep function and sleep progress.
  Interventions: Device: software-delivered CBT-I
- online PE (Active Comparator): Subjects in control group will receive information about insomnia and sleep health education content.
  Interventions: Other: online PE

INTERVENTIONS:
Device: software-delivered CBT-I — The automated software called 'resleep' incorporates all core elements of CBT-I: sleep restriction, stimulus control, cognitive therapy, relaxation techniques, and sleep hygiene and education, tailoring content based on each participant's reported baseline sleep function and sleep progress. The 6-week treatment includes 42 times of intervention.
  Arms: software-delivered CBT-I
Other: online PE — Subjects in the control group will receive non-tailored information about insomnia and sleep health education content using the Wechat Official Account.
  Arms: online PE

SUMMARY:
The goal of this prospective multicenter clinical trial is to evaluate the efficacy and safety of software-delivered cognitive behavioral therapy for insomnia (CBT-I) in Chinese patients with insomnia disorder (ID). The main questions it aims to answer are: (1) whether the software-delivered CBT-I is more effective than an online patient education (online-PE) at improving insomnia. (2) whether the software-delivered CBT-I is safe for treatment of insomnia symptoms.

Participants will be randomized to receive (1) a software-delivered CBT-I using automated software called 'resleep' (one kind of digital device expected to treat insomnia targeted for Chinese patients); (2) online patient education (online-PE) about sleep.

Researchers will compare the efficacy of a software-delivered CBT-I program and an online sleep education control at improving insomnia symptoms and other psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old, no gender limitation;
* Own a mobile-phone, access the Internet, and be skilled in using software;
* Meet the diagnostic criteria of insomnia disorder in the Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition) (DSM-5);
* Insomnia symptoms appear at least 3 nights per week and last for at least 3 months;
* ISI scores ≥ 12 ;
* Volunteer to participate in this experiment and sign a written informed consent.

Exclusion Criteria:

* Generalized Anxiety Disorder Scale-7 (GAD-7) scores ≥ 15;
* Patients Health Questionnaire-9 (PHQ-9) scores ≥ 20;
* Current thoughts of suicide or self-injury (defined as PHQ-9 9th item score ≥ 1);
* Confirmed physical diseases that may affect sleep, such as congestive heart failure, chronic obstructive pulmonary disease acute phase, cardiovascular and cerebrovascular disease acute phase, etc.
* Current diagnosed neurological or mental illness (major depressive disorder, bipolar disorder, epilepsy, schizophrenia, etc.) that may affect sleep;
* Diagnoses of other untreated sleep disorders, such as obstructive sleep apnea, restless leg syndrome (RLS);
* Usual bedtime (when the subject attempts to fall asleep) is earlier than 8 p.m. or later than 2 a.m., or usual waking (arising) time is earlier than 4 a.m. or later than 10 a.m.
* Alcohol or drug abusers (other than nicotine dependence) in the past year;
* Pregnant or lactating women;
* Undergoing systematic psychotherapy within the past 3 months;
* Undergoing other cognitive behavioral therapy for sleep disorders;
* Unstable usage of medication regimens that affect sleep (changes in type, dosage and method of use within the past 1 month);
* Night shift workers, travelers across time zones;
* Subjects who have not responded to previous CBT-I;
* Other conditions deemed unsuitable for clinical trials by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
The Change of Insomnia Severity from Baseline to Follow-up | Baseline, post-intervention, follow-up (3 months after post-intervention)
  The insomnia severity is assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire well validated in insomnia research in multiple patient populations. The change of ISI scores from baseline to follow-up is the primary outcome.

SECONDARY OUTCOMES:
Insomnia Remission | Baseline, post-intervention, follow-up (3 months after post-intervention)
  Insomnia remission was evaluated by a masked assessor using a semi-structured interview.
Insomnia Treatment Response | Baseline, post-intervention, follow-up (3 months after post-intervention)
  Insomnia treatment response was defined by a decrease in ISI by at least 8 points.
Sleep Parameters Assessed by Sleep Diary | Baseline, post-intervention, follow-up (3 months after post-intervention)
  Sleep diaries related parameters include time taken to fall asleep (sleep onset latency), wake after sleep onset, total sleep, total time in bed, and sleep efficiency.
Sleep Quality | Baseline, post-intervention, follow-up (3 months after post-intervention)
  Pittsburgh Sleep Quality Index (PSQI) is used to assess overall sleep quality.
Depression | Baseline, post-intervention, follow-up (3 months after post-intervention)
  Patient Health Questionnaire-9 (PHQ-9) is used to evaluate the severity of depression.
Anxiety | Baseline, post-intervention, follow-up (3 months after post-intervention)
  Generalized Anxiety Disorder Scale-7 (GAD-7) is used to evaluate the severity of anxiety.
Life Quality | Baseline, post-intervention, follow-up (3 months after post-intervention)
  WHOQOL-BREF is used to evaluate the life quality.

OTHER OUTCOMES:
Adverse Events | Baseline, post-intervention, follow-up (3 months after post-intervention)
  Adverse events will be recorded throughout this trial for evaluating the safety of software.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Shenzhen Kangning Hospital, Shenzhen, Guangdong
  - The Second Affiliated Hospital of AFMU, Xi'an, Shaanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No